CLINICAL TRIAL: NCT01796717
Title: Optimizing Dosing Regimen of Piperacillin/Tazobactam, Prolonged Infusion vs. Regular Infusion, Every 6 Hours, for Nosocomial Pneumonia in ICU Caused by Susceptible Pathogens With Higher MIC
Brief Title: Optimizing Dosing Regimen of Piperacillin/Tazobactam for Nosocomial Pneumonia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIH-WDH-201205001
Record Dates: First submitted 2012-08-30; First posted 2013-02-22 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2012-08

CONDITIONS: Nosocomial Pneumonia
Keywords: Piperacillin/tazobactam; MIC
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C Group (Active Comparator): Controlled group will receive piperacillin/tazobactam of 4.5g Q6h, intermittent infusion for 30 minutes
  Interventions: Drug: C Group
- E Group (Experimental): Therapy group will receive piperacillin/tazobactam of 4.5g Q6h, prolonged infusion for 4 hours
  Interventions: Drug: E Group

INTERVENTIONS:
Drug: C Group — Controlled group will receive piperacillin/tazobactam of 4.5g Q6h, intermittent infusion for 30 minutes
  Other Names: nosocomial pneumonia; MIC
  Arms: C Group
Drug: E Group — Therapy group will receive piperacillin/tazobactam of 4.5g Q6h, prolonged infusion for 4 hours
  Other Names: nosocomial pneumonia; MIC
  Arms: E Group

SUMMARY:
1. To observe clinical and bacteriologic responses of different regimens of piperacillin/tazobactam (4.5g q6h, prolonged or intermittent infusion) for treatment of nosocomial pneumonia.
2. To describe the pharmacokinetic profile of piperacillin/tazobactam (4.5g q6h, prolonged or intermittent infusion) in patients with nosocomial pneumonia.
3. To assess the safety profiles of piperacillin/tazobactam 4.5g q6h, prolonged or intermittent infusion in patients with nosocomial pneumonia.

DETAILED DESCRIPTION:
Enrolled patients will be randomized into therapeutic or controlled group. Controlled group will receive piperacillin/tazobactam of 4.5g Q6h, intermittent infusion for 30 minutes. Therapy group will receive piperacillin/tazobactam of 4.5g Q6h, prolonged infusion for 4 hours. The duration is 7-14 days.

Two sets of blood cultures (for aerobic and anaerobic culture) were obtained before the study and post-treatment period if first blood culture is positive. Cultures from the lower respiratory tract infection were obtained before (within 48 h) the study and on the last day of therapy. The lower respiratory tract specimens obtained either by endotracheal aspiration, bronchoalveolar lavage (BAL), a protected brush procedure (PBP) or as sputum were required to show > 25 polymorphonuclear cells and < 10 squamous epithelial cells per field (at 100× magnification).

The plasma concentration of piperacillin and tazobactam will be determined by LC/MS/MS method. The QC samples will also be analyzed simultaneously with each run for the method stability testing, according to the laboratory standard procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 70 years old.
2. Inpatients with nosocomial pneumonia or bacteremia.

   i. Diagnosis of nosocomial pneumonia
   1. Chest radiographic infiltrate that is new or progressive.
   2. At least two or more of the following clinical findings suggesting infection.

      * New onset of fever, oral temperature T>38.3℃ or T<36℃

        * Purulent sputum

          * WBC > 12×10^9/L or <4×10^9/L, or band form >10%

            * PaO2/FIO2<240mmHg

   ii. Diagnosis of bacteremia: Positive blood culture and the isolated bacterial strain are considered to be infection cause.
3. Patients are infected by piperacillin-tazobactam susceptible pathogen with MIC=4, 8 or 16mg/L.

Exclusion Criteria:

1. The patients who received systematic antibacterial treatment more than 48 hours before enrollment and have clinical response.
2. Severe pyemia with hypotension or/and evidences of failure of organic function (shock: systolic pressure < 90mmHg or diastolic pressure < 60mmHg, requiring more than 4 hours of administration of vasopressor(s)；renal impairment: urine volume < 20 ml∕h or < 80 ml∕4h after excluded any other potentials, acute renal failure need dialysis, CLcr<40 mL/min).
3. Documented infection caused by pathogens beyond the antibacterial spectrum of piperacillin/tazobactam.
4. Previously diagnosed condition which tend to mimic or complicate the course and evaluation of the infectious process, e.g. bronchial obstruction, obstructive pneumonia, activate pulmonary malignancy, pulmonary abscess, empyema and active tuberculosis, which might interfere the course of the infectious disease and evaluation of the disease.
5. History of allergy to penicillins.
6. Pregnancy or breast-feeding women.
7. Any conditions investigator considered might increase the risk of patients or interfere study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Extension of the Piperacillin / tazobactam infusion time effect evaluation | 2 weeks
  To observe clinical and bacteriologic responses of different regimens of piperacillin/tazobactam (4.5g q6h, prolonged or intermittent infusion) for treatment of nosocomial pneumonia.

SECONDARY OUTCOMES:
Reducing antibiotic resistance | 2 weeks
  To describe the pharmacokinetic profile of piperacillin/tazobactam (4.5g q6h, prolonged or intermittent infusion) in patients with nosocomial pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Donghao, Chief, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- TianjinCIH, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Roberts JA, Kirkpatrick CM, Roberts MS, Dalley AJ, Lipman J. First-dose and steady-state population pharmacokinetics and pharmacodynamics of piperacillin by continuous or intermittent dosing in critically ill patients with sepsis. Int J Antimicrob Agents. 2010 Feb;35(2):156-63. doi: 10.1016/j.ijantimicag.2009.10.008. Epub 2009 Dec 16. PMID 20018492
- [Background] Wang H, Chen M, Ni Y, Liu Y, Sun H, Yu Y, Yu X, Mei Y, Liu M, Sun Z, Chu Y, Hu Z, Huang X. Antimicrobial resistance among clinical isolates from the Chinese Meropenem Surveillance Study (CMSS), 2003-2008. Int J Antimicrob Agents. 2010 Mar;35(3):227-34. doi: 10.1016/j.ijantimicag.2009.11.010. Epub 2010 Jan 4. PMID 20047820
- [Background] Lorente L, Jimenez A, Martin MM, Iribarren JL, Jimenez JJ, Mora ML. Clinical cure of ventilator-associated pneumonia treated with piperacillin/tazobactam administered by continuous or intermittent infusion. Int J Antimicrob Agents. 2009 May;33(5):464-8. doi: 10.1016/j.ijantimicag.2008.10.025. Epub 2009 Jan 15. PMID 19150225